CLINICAL TRIAL: NCT05326529
Title: To Examine the Effectiveness of Physical Activity, Quality of Life and Hospital Anxiety and Depression Outcomes in Cardiovascular Patients Using Either Traditional, Web-based or a Combined Cardiac Rehabilitation Programme.
Brief Title: Comparison of Traditional, Web-based or a Combined Cardiac Rehabilitation Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chester (Other)
Collaborators: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 290193
Record Dates: First submitted 2022-03-23; First posted 2022-04-13 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2023-05

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiac Rehabilitation; Web-based Cardiac Rehabilitation
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Three way comparison study.
  * Traditional Cardiac Rehabilitation
  * Traditional Cardiac Rehabilitation combined with Web-based Cardiac Rehabilitation
  * Web-based Cardiac Rehabilitation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional Cardiac Rehabilitation (Hospital based programme) (Active Comparator): Traditional Cardiac Rehabilitation will involve 8 hospital-based exercise sessions, and one virtual education day over 8 weeks, supervised by CR health care professionals.
  Interventions: Other: Hospital Based Cardiac Rehabilitation Exercise Classes
- Traditional combined with Web-based Cardiac Rehabilitation (Experimental): Traditional combined with Web-based Cardiac Rehabilitation. Patients will attend 8 hospital-based exercise sessions and one virtual education day over 8-weeks with access to additional web-based (MyHeart app) exercise and educational information.
  Interventions: Other: Hospital Based Cardiac Rehabilitation Exercise Classes; Other: Web-based Cardiac Rehabilitation Exercise Sessions
- Web-based Cardiac Rehabilitation (Experimental): Web-based Cardiac Rehabilitation, using MyHeart app introduced during a pre-CR assessment, will follow an 8-week individualised self-managed platform, allowing contact with the CR health professionals via app messages only (no direct contact for web-based CR).
  Interventions: Other: Web-based Cardiac Rehabilitation Exercise Sessions

INTERVENTIONS:
Other: Hospital Based Cardiac Rehabilitation Exercise Classes — Participants will attend 8 Hospital based CR exercise sessions. QOL and Hospital anxiety and Depression scores through questionnaires and incremental Shuttle Walk tests will be carried out pre and post intervention.
  Arms: Traditional Cardiac Rehabilitation (Hospital based programme); Traditional combined with Web-based Cardiac Rehabilitation
Other: Web-based Cardiac Rehabilitation Exercise Sessions — Participants will complete 8 weeks of Web-based CR exercise sessions using the MyHeart app. QOL and Hospital anxiety and Depression scores through questionnaires and incremental Shuttle Walk tests will be carried out pre and post intervention.
  Arms: Traditional combined with Web-based Cardiac Rehabilitation; Web-based Cardiac Rehabilitation

SUMMARY:
The study explores the different modes of Cardiac Rehabilitation delivery including the use of a web-based programme. Cardiac Rehabilitation provides a structured, comprehensive programme, proven to reduce cardiovascular mortality and improve overall Quality of Life. However, as uptake remains relatively low with only 50% attending, exploring the benefits of offering a menu of programme options may allow greater patient choice and accessibility, meeting individual needs.

This study aims to compare how effective Cardiac Rehabilitation Programmes are on improving cardiovascular patients physical and mental wellbeing using a web-based compared with traditional cardiac rehab programmes in the hospital or through a combination of both.

DETAILED DESCRIPTION:
This 8-week study, aims to compare quality of life (QOL), hospital anxiety and depression scores (HADs) and physical activity outcomes in web-based Cardiac Rehabilitation (CR), web-based CR combined with traditional CR (TCR) and TCR in patients with coronary heart disease (CHD).

The Web-based option will include the use of the MyHeart application.

Participants eligible for the study will include low-moderate cardiovascular patients (heart attack, stents or heart surgery) within 3-6 weeks post discharge. Participants will be involved in hospital or virtual exercise and educational sessions with the support of CR specialists. Primary outcomes will be measured through questionnaires and an incremental treadmill walking test.

To our knowledge, this would be the first study to compare all three groups, as combined CR (web-based alongside traditional CR) has not yet been evaluated. Additionally, the investigators currently work within the CR setting at Burton Hospital, and this study will be conducted within our current Hospital CR service. The outcomes will be applicable and relevant to future clinical practice.

As the UK's 50% uptake to CR remains poor, falling below the 85% national uptake recommendations, a CR menu-based approach, offering hospital or home-based programmes is recommended to encourage uptake, improve QOL and clinical outcomes.

Furthermore, as COVID-19 has enforced a web-based CR approach, further research to explore uptake, physical and psychological outcomes to benefit cardiovascular patients is paramount for current and future CR delivery.

This study will explore a menu of options recommended for CR.

ELIGIBILITY:
Inclusion Criteria:

* Low-moderate risk patients (low-mod Ejection Fraction (EF) (>40%), including clinically stable Myocardial Infarction (MI), Percutaneous Coronary Intervention (PCI), Coronary Artery Bypass Grafts (CABG) patients.
* Acute patients, in-hospital patients (phase 3 rehab) to reflect true clinical representation.
* Combination of male and female, as previous studies are predominately male.
* Low-moderate Anxiety and depression scores (<11)
* Achieve Level 4 (180metres, 5.1METs) on the Incremental Shuttle Walking Test
* Internet and device access.

Exclusion Criteria:

* <40% EF
* High risk Heart Failure patients
* Co-morbidities preventing exercise
* No internet access
* Unstable angina
* Language barrier (English only, due to app)
* Clinically depressed anxiety or depression scores (>11)
* Incremental Shuttle Walk Test <Level 4 (180metres, 5.1METs)

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Morris, Study Director — University of Chester
Locations (1):
- University of Derby and Burton NHS Foundation Trust, Burton-on-Trent, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brough C, Boyce S, Houchen-Wolloff L, Sewell L, Singh S. Evaluating the interactive web-based program, activate your heart, for cardiac rehabilitation patients: a pilot study. J Med Internet Res. 2014 Oct 29;16(10):e242. doi: 10.2196/jmir.3027. PMID 25359204

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started 7/7/22 - ended 28/2/23 Hospital based programme - Queens hospital Burton, UK - Cardiac Rehabilitation Department
Period: Overall Study
Arm/Group | Traditional Cardiac Rehabilitation (Hospital Based Programme) | Traditional Combined With Web-based Cardiac Rehabilitation | Web-based Cardiac Rehabilitation
Started | 19 | 19 | 19
Completed | 19 | 18 | 17
Not Completed | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Cardiac Rehabilitation (Hospital Based Programme) | Traditional Combined With Web-based Cardiac Rehabilitation | Web-based Cardiac Rehabilitation | Total
Number analyzed (Participants) | 19 | 19 | 19 | 57
Age, Customized [Number; unit: participants] — 50-70 years old patients
  participants
    Age 50- 70 years | 19 | 19 | 19 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 2 | 11
  Male | 13 | 16 | 17 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 19 | 19 | 19 | 57

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Energy Expenditure (Measured in METs Using the BACPR Conversion Chart) and After 8 Weeks of Intervention.
Description: An Incremental Shuttle Walk test will be performed to determine the Metabolic equivalent achieved at each level. Metabolic Equivalent (1 MET) is defined as the amount of energy required to serve the body's energy needs. This will range from 1 METs = lowest energy requirement to 10.9 METs highest energy requirement for completing the test. Walking at a slower pace requires a lower level of energy expenditure and is therefore considered a light-intensity activity, walking at a faster pace requires a higher energy expenditure and is therefore considered a higher-intensity activity. The higher the score the better the outcome for the participant as they are able to work at a higher level of exercise and thus an increase functional capacity which equates to a reduction in risk of mortality.
Time Frame: The Walk Test will be completed pre and post intervention (8 weeks apart)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Traditional Cardiac Rehabilitation (Hospital Based Programme) | Traditional Combined With Web-based Cardiac Rehabilitation | Web-based Cardiac Rehabilitation
Number analyzed (Participants) | 19 | 18 | 17
score on a scale
  Pre intervention | 5.9 [5.5 to 6.4] | 5.8 [5.4 to 6.2] | 5.6 [5.2 to 6.0]
  Post Intervention | 7.4 [6.9 to 7.9] | 7.3 [6.9 to 7.7] | 6.5 [6.1 to 7.0]

2. Secondary Outcome: Psychological Outcome - Hospital Anxiety and Depression Score Pre and Post Intervention
Description: This will be evaluated through participants completing a Hospital Anxiety and Depression questionnaire. Scoring range: 0-7 = normal range, 8-10 = borderline abnormal,11-21 abnormal and treatment is indicated. The questionnaire comprises of 7 questions for Anxiety and 7 for Depression with a total score for each ranging from 1-21. The scores will be reported separately for Anxiety and depression. The higher the score the worse the outcome for the participant as this indicates a higher level of either anxiety or depression.
Time Frame: Questionnaires will be given to the patient to complete pre and post intervention. (8 weeks apart)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Cardiac Rehabilitation (Hospital Based Programme) | Traditional Combined With Web-based Cardiac Rehabilitation | Web-based Cardiac Rehabilitation
Number analyzed (Participants) | 19 | 18 | 17
score on a scale
  Pre Intervention (Anxiety Score) | 4.95 (3.1) | 4.56 (3.05) | 5.65 (3.25)
  Post Intervention (Anxiety Score) | 3.68 (2.45) | 4.00 (3.77) | 4.53 (2.98)
  Pre Intervention (Depression Score) | 4.53 (3.58) | 3.28 (2.42) | 4.59 (3.22)
  Post Intervention (Depression Score) | 3.16 (2.47) | 2.44 (2.09) | 3.94 (3.03)

3. Secondary Outcome: Psychological Status at Baseline (Using the Dartmouth Coop Questionnaire) and After 8 Weeks of Intervention.
Description: This will be evaluated through participants completing a questionnaire consisting of questions measuring health status, physical fitness, feelings, daily activities, social activities, change in health status, current overall health perceptions and bodily pain. Each question gives 5 response options, 1= very good, 2= good, 3= Moderate, 4=Bad, 5= Very Bad. Minimum score = 9, maximum score 45. Total score gives a profile of health status i.e, higher total score = poor health status. The scores will be evaluated at baseline and after 8 weeks of intervention. The score should be lower after 8 weeks to a reflect an improvement in overall health status.
Time Frame: Questionnaires will be given to the patient to complete pre and post intervention. (8 weeks apart)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Cardiac Rehabilitation (Hospital Based Programme) | Traditional Combined With Web-based Cardiac Rehabilitation | Web-based Cardiac Rehabilitation
Number analyzed (Participants) | 19 | 18 | 17
score on a scale
  Pre Intervention | 21.9 (5.63) | 20.1 (5.01) | 21.35 (5.38)
  Post Intervention | 16.4 (3.57) | 15.7 (2.63) | 17.41 (4.50)

4. Secondary Outcome: Heart Rate Walking Speed Index at Baseline and After 8 Weeks of Intervention
Description: An Incremental Shuttle Walk test will be performed to evaluate functional capacity and determine what percentage of predicted heart rate the participant has achieved at each level of the walk test. The maximum Heart Rate achieved at the end of the walk test will then be converted to walking speed index (HRWSI). This will be converted using the BACPR HRWSI table which looks at the number of heart beats for every 10 meters walked when completing a standardised walking test. HRWSI is calculated by dividing Heart rate by the walking speed (meters per minute) multiplied by 10 to give heart beats per minute walked. Possible score ranges are 3-90 (heart beats per 10 meters). If heart rate has decreased at any given point of the walking test compared with the baseline test, this represents an increase in aerobic fitness.
Time Frame: The Walk Test will be completed pre and post intervention (8 weeks apart)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Traditional Cardiac Rehabilitation (Hospital Based Programme) | Traditional Combined With Web-based Cardiac Rehabilitation | Web-based Cardiac Rehabilitation
Number analyzed (Participants) | 19 | 18 | 17
score on a scale
  Pre Intervention | 11.3 [10.2 to 12.5] | 11.3 [10.5 to 12.1] | 12.2 [11.1 to 13.3]
  Post Intervention | 10.2 [9.3 to 11.1] | 10.2 [9.6 to 10.8] | 10.9 [9.8 to 12.2]

ADVERSE EVENTS:
Time Frame: 8 weeks (duration of the exercise component part of the study)
Arm/Group | Traditional Cardiac Rehabilitation (Hospital Based Programme) | Traditional Combined With Web-based Cardiac Rehabilitation | Web-based Cardiac Rehabilitation
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT05326529/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT05326529/ICF_001.pdf